CLINICAL TRIAL: NCT00740376
Title: A Prospective, Comparative, Randomized, Double Blind, Multi-center Study of the Uniglide™ Mobile Bearing Unicondylar Knee System vs. Uniglide™ Fixed Bearing Unicondylar Knee System
Brief Title: Uniglide™ Mobile Bearing Unicondylar Knee System vs the Uniglide™ Fixed Bearing Unicondylar Knee System
Acronym: MBK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Uniglide MBK
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-05

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Uniglide Mobile Bearing (Experimental): Uniglide Mobile Bearing Unicondylar Knee System (MBK)
  Interventions: Device: Uniglide Mobile Bearing Unicondylar Knee System
- Uniglide Fixed Bearing (Active Comparator): Uniglide Fixed Bearing Unicondylar Knee System (FBK)
  Interventions: Device: Uniglide Fixed Bearing Unicondylar Knee System

INTERVENTIONS:
Device: Uniglide Mobile Bearing Unicondylar Knee System — Uniglide Mobile Bearing Knee System includes a femoral component made of cobalt chromium molybdenum (CoCrMo)that articulates with a mobile bearing tibial construct comprised of a cobalt chromium molybdenum (CoCrMo)tibial base plate and ultra high molecular weight polyethylene (UHMWPE) meniscal insert. The femoral component has been cleared as part of the fixed bearing version in K050764. The investigational portion of this device is the mobile bearing tibial construct (tibial tray and meniscal insert).
  Other Names: unicondylar knee; unicompartmental knee; partial knee
  Arms: Uniglide Mobile Bearing
Device: Uniglide Fixed Bearing Unicondylar Knee System — Uniglide Fixed Bearing Knee System includes a femoral component made of cobalt chromium molybdenum (CoCrMo) that articulates with a one piece ultra high molecular weight polyethylene (UHMWPE) tibial bearing (K050764).
  Other Names: unicondylar knee; unicompartmental knee; partial knee
  Arms: Uniglide Fixed Bearing

SUMMARY:
The purpose of this study is to demonstrate that the Uniglide™ Mobile Bearing Unicondylar Knee System (investigational device)is not inferior when compared to the Uniglide™ Fixed Bearing Unicondylar Knee System (control device currently cleared) as measured by the Composite Clinical Success (CCS) endpoint.

DETAILED DESCRIPTION:
Arthritic knees are the most common cause of long-term disability resulting in decreased mobility and increased pain. After other treatments for pain relief and return to activities of daily living fail, knee joint replacement is often the best option and unicompartmental knee arthroplasty was introduced as an appropriate treatment for management of osteoarthritis when disease effects only a portion of the knee joint. This study is a prospective, comparative, randomized, double blind (patient and post-operative evaluator), multi-center clinical study under a common protocol to determine the safety and effectiveness of the Uniglide Unicondylar Mobile Bearing knee implant system.

ELIGIBILITY:
Inclusion Criteria:

* skeletally mature
* need to obtain pain relief and improved function
* moderate or severe pain with either walking or at rest on the Hospital for Special Surgery Score
* preoperative medial tibiofemoral joint space narrowing on x-rays (Kellgren Lawrence grade 3 or 4)
* preoperative Hospital for Special Surgery Knee Evaluation total score of < 69
* preoperative arc of motion of > 90o in the affected knee
* diagnosed with osteoarthritis in the medial compartment of the knee and non-surgical treatment options have failed to provide relief for symptoms
* able to understand this clinical trial, co-operate with study procedures, and are willing to return to the clinic, and/or hospital for all the required post-operative follow-ups
* able to give and have given voluntary, written informed patient consent to participate in this clinical investigation and have provided Authorization for Release of Personal Health Information (HIPAA) for the purpose of this clinical study
* willing to be randomized with either of the devices used in the clinical trial as determined by the randomization schedule

Exclusion Criteria:

* neurological disorders which may interfere or adversely affect gait or weight bearing (e.g., muscular dystrophy, multiple sclerosis)
* a nutritional problem (protein, calorie, or vitamin/mineral deficiency) that may impair wound healing mechanisms
* a diagnosed systemic disease that would affect their welfare or the overall outcome of study (i.e. Paget's disease, renal osteodystrophy)
* immunologically suppressed
* on chronic corticosteroid or non-steroidal anti-inflammatory therapy
* with Charcot's disease
* with metabolic disorders (e.g. osteomalacia), which may impair bone formation
* with distant foci of infections, which may spread to the implant site
* have presence of vascular insufficiency, muscular atrophy and neuromuscular disease
* have diagnosed osteoporosis as evidenced on a DEXA scan (within the last 12 months)
* ave diagnosed rheumatoid arthritis or other forms of inflammatory joint disease
* have diagnosed avascular necrosis
* with malunion, arthrodesis or severe dysplasia in the affected limb
* with rapid joint destruction, marked bone loss or bone resorption in the affected knee apparent on x-ray
* have incomplete or deficient soft tissue surrounding the affected knee
* have infection, sepsis or osteomyelitis in the affected knee
* have had revision of previously failed prosthesis, failed upper tibial osteotomy or post traumatic arthritis after tibial plateau fracture in the affected knee
* with a fixed varus deformity (not passively correctable) of greater than 15 degrees and a flexion deformity greater than 15 degrees in the affected knee
* with insufficient collateral, anterior or posterior cruciate ligaments in the affected knee, which would preclude stability of the device
* with disease or damage to the lateral compartment of the affected knee (Outerbridge classification II, III, or IV)
* with a Body Mass Index > 36
* with a sensitivity to device material
* Females who are pregnant
* prisoners,known drug or alcohol abuser, smoker, or have a psychological disorder
* Based upon intra-operative assessment, cartilage and bone erosions involving more than the anterior and middle parts of the medial compartment. The posterior part of the medial compartment and the lateral compartment having cartilage of less than normal thickness. (as assessed using the Outerbridge Classification system).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Fleming, Study Director — Corin Ltd
Locations (6):
- United States (6):
  - S.T.A.R. Orthopaedics, Inc., La Quinta, California
  - Orthopaedic Associates of West Florida, Clearwater, Florida
  - Bluegrass Orthopaedics and Hand Care, Lexington, Kentucky
  - Texas Orthopedic Specialists, Bedford, Texas
  - Memorial Bone & Joint, Houston, Texas
  - Texas Center for Joint Replacement, Plano, Texas

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Implants
Groups:
- Uniglide Mobile Bearing Unicondylar Knee System (MBK): Uniglide Mobile Bearing Unicondylar Knee System (MBK)
  Uniglide Mobile Bearing Unicondylar Knee System: Uniglide Mobile Bearing Knee System includes a femoral component made of cobalt chromium molybdenum (CoCrMo) that articulates with a mobile bearing tibial construct comprised of a cobalt chromium molybdenum (CoCrMo) tibial base plate and ultra high molecular weight polyethylene (UHMWPE) meniscal insert. The femoral component has been cleared as part of the fixed bearing version in K050764. The investigational portion of this device is the mobile bearing tibial construct (tibial tray and meniscal insert).
- Uniglide Fixed Bearing Unicondylar Knee System (FBK): Uniglide Fixed Bearing Unicondylar Knee System (FBK)
  Uniglide Fixed Bearing Unicondylar Knee System: Uniglide Fixed Bearing Knee System includes a femoral component made of cobalt chromium molybdenum (CoCrMo) that articulates with a one piece ultra high molecular weight polyethylene (UHMWPE) tibial bearing (K050764).
Period: Overall Study
Arm/Group | Uniglide Mobile Bearing Unicondylar Knee System (MBK) | Uniglide Fixed Bearing Unicondylar Knee System (FBK)
Started | 22; 26 Implants | 15; 21 Implants
Completed | 19; 22 Implants | 12; 18 Implants
Not Completed | 3; 4 Implants | 3; 3 Implants

BASELINE CHARACTERISTICS:
Units Other Than Participants: Implants
Groups:
- Total: Total of all reporting groups
Arm/Group | Uniglide Mobile Bearing Unicondylar Knee System (MBK) | Uniglide Fixed Bearing Unicondylar Knee System (FBK) | Total
Number analyzed (Participants) | 22 | 15 | 37
Number analyzed (Implants) | 26 | 21 | 47
Age, Continuous [Mean (Full Range); unit: years] | 60.42 [48 to 71] | 57.48 [43 to 77] | 58.95 [43 to 77]
Sex: Female, Male [Count of Units; unit: Implants]
  Female | 18 | 7 | 25
  Male | 8 | 14 | 22
Region of Enrollment [Number; unit: Implants]
  United States | 26 | 21 | 47

OUTCOME MEASURES:

1. Primary Outcome: The Number of Implants Which Achieve Composite Clinical Success (CCS) at Month 24.
Description: CCS success criteria includes the following:
  Hospital for Special Surgery (HSS) success: ≥ 70 and; If preop HSS between 60-69, HSS ≥ 70 plus a min 10 point improvement;
  No radiographic failure: No radiolucent lines >1mm in >50% of zones around any component; No progressive radiolucencies; No radiographic evidence of implant subsidence (vertical displacement) > 2mm of any component; No radiographic evidence of aseptic implant loosening, i.e. no changes in angular orientations > 2 degrees;
  No removal, replacement, or revision (including planned removal, replacement, or revision) of any component (including the bearing) on or before day 730 following initial surgery.
Time Frame: Month 24 postoperative
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Uniglide Mobile Bearing Unicondylar Knee System (MBK) | Uniglide Fixed Bearing Unicondylar Knee System (FBK)
Number analyzed (Participants) | 19 | 12
Number analyzed (Implants) | 22 | 18
Implants | 17 | 15

2. Secondary Outcome: American Knee Society Score (AKSS) (Total, Pain & Function Scores)
Description: American Knee Society Score (AKSS) Total Score - Range: 0 (worst) - 100 (best) Pain Score - Range: 0 (worst) - 50 (best) Function Score - Range: 0 (worst) - 100 (best)
Time Frame: Month 24 postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Implants
Arm/Group | Uniglide Mobile Bearing Unicondylar Knee System (MBK) | Uniglide Fixed Bearing Unicondylar Knee System (FBK)
Number analyzed (Participants) | 17 | 13
Number analyzed (Implants) | 20 | 19
score on a scale
  Mean Pain Score | 48.00 (6.77) | 42.63 (10.32)
  Mean Function Score | 95.50 (10.50) | 94.74 (11.72)
  Mean Total Score | 94.53 (8.46) | 89.58 (12.87)

3. Secondary Outcome: Hospital for Special Surgery (HSS) Score (Total, Pain & Function Scores)
Description: HSS (total): range 0 (worst) - 100 (best) HSS (pain): range 0 (worst) - 30 (best) HSS (function): range 0 (worst) - 22 (best)
Time Frame: Month 24 postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Implants
Arm/Group | Uniglide Mobile Bearing Unicondylar Knee System (MBK) | Uniglide Fixed Bearing Unicondylar Knee System (FBK)
Number analyzed (Participants) | 17 | 13
Number analyzed (Implants) | 20 | 19
score on a scale
  Mean Total Score | 95.25 (5.31) | 93.63 (6.18)
  Mean Pain Score | 29.25 (2.45) | 28.16 (3.80)
  Mean Function Score | 21.30 (1.78) | 20.79 (1.51)

4. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS) (Pain, Symptoms, Activities of Daily Living, Sports/Rec & Quality of Life Scores)
Description: Knee injury and Osteoarthritis Outcome Score (pain): 0 (worst) - 100 (best) Knee injury and Osteoarthritis Outcome Score (symptoms): 0 (worst) - 100 (best) Knee injury and Osteoarthritis Outcome Score (activities of daily living (ADL)): 0 (worst) - 100 (best) Knee injury and Osteoarthritis Outcome Score (sport/rec): 0 (worst) - 100 (best) Knee injury and Osteoarthritis Outcome Score (quality of life (QOL)): 0 (worst) - 100 (best)
  Knee injury and Osteoarthritis Outcome Score (sport and recreation): 0 (worst) - 100 (best)
  Knee injury and Osteoarthritis Outcome Score (quality of life): 0 (worst) - 100 (best)
Time Frame: Month 24 postoperative
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Implants
Arm/Group | Uniglide Mobile Bearing Unicondylar Knee System (MBK) | Uniglide Fixed Bearing Unicondylar Knee System (FBK)
Number analyzed (Participants) | 17 | 13
Number analyzed (Implants) | 17 | 12
score on a scale
  Mean Pain Score | 91.35 (11.15) | 92.00 (9.71)
  Mean Symptoms Score | 63.82 (13.87) | 66.73 (15.54)
  Mean ADL Score | 93.65 (10.21) | 92.67 (9.80)
  Mean Sport/Rec Score | 77.94 (21.22) | 78.67 (21.17)
  Mean QOL Score | 83.94 (15.11) | 84.27 (13.26)

5. Secondary Outcome: Survival Rate Using Kaplan-Meier Survival Curves
Description: Kaplan-Meier survival curves will be plotted for All Enrolled investigational devices and All Enrolled control devices on the same graph to facilitate graphical comparisons of survivorship over time.
Time Frame: Month 24 postoperative
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Uniglide Mobile Bearing Unicondylar Knee System (MBK) | Uniglide Fixed Bearing Unicondylar Knee System (FBK)
Number analyzed (Participants) | 22 | 15
Number analyzed (Implants) | 26 | 21
Implants | 24 | 21

6. Secondary Outcome: Number of Implants With Any Device-related Complications
Time Frame: Month 24 postoperative
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Uniglide Mobile Bearing Unicondylar Knee System (MBK) | Uniglide Fixed Bearing Unicondylar Knee System (FBK)
Number analyzed (Participants) | 22 | 15
Number analyzed (Implants) | 26 | 21
Implants | 3 | 0

7. Secondary Outcome: The Number of Implants With Any Radiographic Findings at Month 24 Post Operatively
Description: For both the Tibial & Femoral Components the following were recorded:
  Implant Subsidence > 2mm (recorded for the tibial component only) Implant Loosening > 2deg Radiolucent Line (RLL) in >50% zones Progressive RLL Osteolysis ≥ 5mm
Time Frame: Month 24 postoperative
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Uniglide Mobile Bearing Unicondylar Knee System (MBK) | Uniglide Fixed Bearing Unicondylar Knee System (FBK)
Number analyzed (Participants) | 17 | 12
Number analyzed (Implants) | 20 | 18
Implants
  Tibial Implant Subsidence | 0 | 0
  Tibial Implant Loosening | 0 | 0
  Tibial RLL | 1 | 1
  Tibial Progressive RLL | 3 | 1
  Tibial Osteolysis | 1 | 0
  Femoral Implant Loosening | 0 | 0
  Femoral RLL | 0 | 1
  Femoral Progressive RL | 0 | 1
  Femoral Osteolysis | 0 | 0

ADVERSE EVENTS:
Arm/Group | Uniglide Mobile Bearing Unicondylar Knee System (MBK) | Uniglide Fixed Bearing Unicondylar Knee System (FBK)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/15
Serious Adverse Events (participants affected / at risk) | 6/22 | 7/15
Other Adverse Events (participants affected / at risk) | 20/22 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Uniglide Mobile Bearing Unicondylar Knee System (MBK) (N=22) | Uniglide Fixed Bearing Unicondylar Knee System (FBK) (N=15)
Chronic lymphocytic leukaemia anemia (Blood and lymphatic system disorders) | 1 | 0
Chronic lymphocytic leukaemia progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Contralateral hip arthrotomy for loose body removal (Surgical and medical procedures) | 1 | 0
Contralateral UKR (Surgical and medical procedures) | 1 | 0/5
Contralateral TKR (Surgical and medical procedures) | 2 | 0
Closed reduction percutaneous screw fixation of ipsilateral subcapital femoral neck fracture (Surgical and medical procedures) | 1 | 0
Revision for meniscal bearing dislocation (Surgical and medical procedures) | 1 | 0
Revision for periprosthetic fracture (Surgical and medical procedures) | 1 | 0
Carpal tunnel release surgery (Surgical and medical procedures) | 0 | 1
Contralateral knee hematoma drainage (Surgical and medical procedures) | 0 | 1
Contralateral knee traumatic wound dehiscence (Surgical and medical procedures) | 0 | 1
Gastrointestinal polyp removal (Surgical and medical procedures) | 0 | 1
Knee hematoma drainage (operative side) (Surgical and medical procedures) | 0 | 1
Lumbago (Musculoskeletal and connective tissue disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
Traumatic knee-wound dehiscence (operative side) (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Uniglide Mobile Bearing Unicondylar Knee System (MBK) (N=22) | Uniglide Fixed Bearing Unicondylar Knee System (FBK) (N=15)
Achiness and sensitivity both knees (Skin and subcutaneous tissue disorders) | 1 | 0
Acute post-op blood loss anemia (Injury, poisoning and procedural complications) | 3 | 1
Ankle swelling (Injury, poisoning and procedural complications) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 4
Contralateral hallux rigidus surgery (Surgical and medical procedures) | 1 | 0
Contralateral hip OA (Musculoskeletal and connective tissue disorders) | 1 | 0
Contralateral hip pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Contralateral knee crepitus (Musculoskeletal and connective tissue disorders) | 1 | 0
Contralateral knee OA (Musculoskeletal and connective tissue disorders) | 1 | 1
Contralateral knee pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Contralateral meniscus tear (Injury, poisoning and procedural complications) | 1 | 0
Contralateral twisted knee (Injury, poisoning and procedural complications) | 1 | 0
Drainage from incision (Surgical and medical procedures) | 1 | 0
Fever (Infections and infestations) | 2 | 0
Gas pain (Gastrointestinal disorders) | 1 | 0
Heartburn (Gastrointestinal disorders) | 1 | 1
Heterotopic ossification (operative side) (Musculoskeletal and connective tissue disorders) | 1 | 0
Indigestion (Gastrointestinal disorders) | 1 | 0
Itching (Skin and subcutaneous tissue disorders) | 2 | 2
Knee and ankle swelling (operative side) (Musculoskeletal and connective tissue disorders) | 1 | 0
Knee crepitus (operative side) (Musculoskeletal and connective tissue disorders) | 1 | 0
Knee pain (operative side) (Musculoskeletal and connective tissue disorders) | 2 | 2
Knee swelling and discomfort (operative side) (Injury, poisoning and procedural complications) | 1 | 0
Left elbow and head bruising (Injury, poisoning and procedural complications) | 1 | 0
Muscle spasm (Musculoskeletal and connective tissue disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 7 | 7
Nausea and vomiting (Gastrointestinal disorders) | 4 | 1
Numbness and tingling (Nervous system disorders) | 1 | 0
Off-label drill bit breakage during surgery (Injury, poisoning and procedural complications) | 1 | 0
Pes anserine bursitis (operative side) (Musculoskeletal and connective tissue disorders) | 2 | 1
Post-fall bruised knee (operative side) (Injury, poisoning and procedural complications) | 1 | 1
Post-fall contralateral knee pain (Injury, poisoning and procedural complications) | 1 | 0
Post-fall knee contusion (operative side) (Injury, poisoning and procedural complications) | 1 | 0
Post-fall knee pain (operative side) (Injury, poisoning and procedural complications) | 3 | 1
Productive cough with yellow discharge (Infections and infestations) | 1 | 0
Rash on back and chest (Skin and subcutaneous tissue disorders) | 1 | 0
Skin cancer (left shin) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sleeplessness (General disorders) | 3 | 0
Sore throat (Infections and infestations) | 1 | 0
Total hysterectomy (Reproductive system and breast disorders) | 1 | 0
Twisted knee (operative side) (Injury, poisoning and procedural complications) | 1 | 0
Uncharacteristic pain (operative side) (Musculoskeletal and connective tissue disorders) | 1 | 1
All over general itching (Skin and subcutaneous tissue disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
C-6 calcification (Musculoskeletal and connective tissue disorders) | 0 | 1
Contralateral knee arthroscopy (Surgical and medical procedures) | 0 | 1
Contralateral pes anserine bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Early degenerative changes in lumbar spine (Musculoskeletal and connective tissue disorders) | 0 | 1
Elbow pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Elevated blood pressure (Cardiac disorders) | 0 | 1
Fractured foot (Injury, poisoning and procedural complications) | 0 | 1
Hypertension (Cardiac disorders) | 0 | 1
Insomnia (General disorders) | 0 | 4
Ipsilateral hip bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Knee arthroscopy (operative side) (Surgical and medical procedures) | 0 | 1
Knee locking (operative side) (Musculoskeletal and connective tissue disorders) | 0 | 1
Lethargy (General disorders) | 0 | 1
Mole removal (Surgical and medical procedures) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nausea and vomiting (Gastrointestinal disorders) | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 1
Occasional contralateral intertrochanteric hip pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Post-fall bruised contralateral knee (Injury, poisoning and procedural complications) | 0 | 1
Post-op nausea (Injury, poisoning and procedural complications) | 0 | 1
Progression of OA (Musculoskeletal and connective tissue disorders) | 0 | 1
Vomiting and diarrhea (Gastrointestinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days